CLINICAL TRIAL: NCT01530932
Title: Immune Activation, Hypoxia and Vasoreaction in Sepsis of Pulmonary Versus Abdominal Origin
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Timo Sturm, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2011-411M-MA
Record Dates: First submitted 2011-11-09; First posted 2012-02-10 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Sepsis
Keywords: sepsis; tissue oxygenation; tissue perfusion; immune reaction
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sepsis remains a common entity in critical care patients with remarkable mortality. Pulmonary and abdominal infections (with subsequent sepsis) are the most common in the ICU. Despite extended research activities, no differences in patient outcome or organ dysfunction were revealed.

Sepsis is a complex immune reaction phenomenon based on unbalanced activation and suppression. In addition to changes of cytokine levels and immune cell activity, underlying genetic reactions are present. For instance, expression of miRNA (as a potential important step of immune cell activation) is likely changed during systemic and local immune reactions.

The aim of this study is to perform a detailed assay of immune cell activation, to investigate the levels of pro- and antiinflammatory cytokines and the various expression of miRNA depending on the origin of infection in the two most common sides. This means in ICU patients with early pulmonary or abdominal sepsis as well as in healthy controls. Additionally, clinical parameters of organ function, current infection markers as CRP and procalcitonin, cardiovascular function and heart rate variability will be assessed. Parameters of local tissue perfusion in a dynamic testing during forearm ischemia and plasma adenosine concentration will be measured.

ELIGIBILITY:
Inclusion Criteria:

* sepsis (according to the criteria of the International Sepsis Definition Conference)

Exclusion Criteria:

* pregnancy
* malignancy
* corticoid therapy
* organ transplantation
* renal insufficiency with HD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis of pulmonary or abdominal origin with admission to the ICU in the first 48 hours of sepsis onset
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Sturm T, Leiblein J, Clauss C, Erles E, Thiel M. Bedside determination of microcirculatory oxygen delivery and uptake: a prospective observational clinical study for proof of principle. Sci Rep. 2021 Dec 31;11(1):24516. doi: 10.1038/s41598-021-03922-4. PMID 34972827
- [Derived] Sturm T, Leiblein J, Schneider-Lindner V, Kirschning T, Thiel M. Association of Microcirculation, Macrocirculation, and Severity of Illness in Septic Shock: A Prospective Observational Study to Identify Microcirculatory Targets Potentially Suitable for Guidance of Hemodynamic Therapy. J Intensive Care Med. 2018 Apr;33(4):256-266. doi: 10.1177/0885066616671689. Epub 2016 Sep 29. PMID 27686326